CLINICAL TRIAL: NCT01037114
Title: An Open Single Centre Study to Evaluate the Long-term Antibody Persistence and Immune Memory Between 16 and 20 Years After the Primary Study HAB-032 (208127/022) in Which Healthy Adults Were Vaccinated With Twinrix Adult Following a Three-dose Schedule.
Brief Title: Long-term Persistence Study in Healthy Adults Previously Vaccinated With Twinrix Adult
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112266
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis A; Hepatitis B
Keywords: Hepatitis A and hepatitis B
MeSH Terms: conditions — Hepatitis A; Hepatitis B | interventions — Blood Specimen Collection; Engerix-B; Hepatitis A Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Twinrix Group (Experimental): Subjects who received 2 doses of Twinrix (lot A, B or C) in the primary study.
  As lot to lot consistency was assessed during the primary study, the 3 groups (lot A, B or C) were pooled into the Twinrix Group for data analyses during the first long-term follow-up NCT00289718 and this long-term follow-up.
  A challenge dose of the Havrix or Engerix-B vaccines can be administered in this study based on serology results at each time point.
  Interventions: Procedure: Blood sampling; Biological: Engerix-B; Biological: Havrix

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling at Year 16, 17, 18, 19 and 20 and at the time of challenge dose administration and 14 days and one month after challenge dose administration (if challenge dose needed).
Biological: Engerix-B — Engerix-B will be administered to subjects who are not seroprotected against hepatitis B.
Biological: Havrix — Havrix will be administered to subjects who are seronegative for anti-HAV antibodies.

SUMMARY:
This study will evaluate the persistence of the immune response to HAV (hepatitis A virus) antigens and HBs (hepatitis B surface) antigens in healthy adults previously vaccinated with Twinrix Adult in the primary study, HAB-032 (208127/022). The subjects will be invited for blood sampling 16, 17, 18, 19 and 20 years after the primary vaccination to evaluate the antibody persistence. For subjects in whom low circulating antibodies are detected, the presence of immune memory against hepatitis A & B antigens will be investigated by the administration of a challenge dose of the appropriate vaccine (Havrix and/or Engerix-B) at the next planned visit.

No new subjects will be recruited during this study.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at entry into each of the long-term follow-up visits:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female who received the complete primary vaccination course in the primary study 208127/022.
* Written informed consent obtained from the subject.

All subjects must satisfy the following criteria at entry into the challenge dose phase:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female who received the complete primary vaccination course in the primary study 208127/022.
* Written informed consent obtained from the subject.
* Subjects who participated in the LTFU phase of the 208127/022 study and for whom the antibody concentrations were below the cut-off at the last available follow-up time-point.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception for two months after the administration of the challenge dose.

Exclusion Criteria:

The following criteria should be checked before entry into each of the long-term follow-up visits. If any exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product within 30 days prior to blood sampling.
* Administration of a hepatitis A, hepatitis B or combined hepatitis A and B vaccine outside the study procedures, since the primary study 208127/022.
* History of hepatitis A or hepatitis B infection since the primary study 208127/022.
* Administration of hepatitis A or hepatitis B immunoglobulins and/or any blood products within three months prior to blood sampling.

The following criteria should be checked before the challenge dose is administered. If any apply, the subject must not be included in the challenge dose phase:

* Use of any investigational or non-registered product within 30 days prior to study start or planned use during the study.
* Administration of a hepatitis A, hepatitis B or combined hepatitis A and B vaccine between the last LTFU visit and the challenge dose visit.
* History of hepatitis A or hepatitis B infection between the last LTFU visit and the challenge dose visit.
* History of anaphylactic reactions following the administration of vaccines.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01-27 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Agrawal A, Kolhapure S, Andani A, Ota MOC, Badur S, Karkada N, Mitra M. Long-Term Persistence of Antibody Response with Two Doses of Inactivated Hepatitis A Vaccine in Children. Infect Dis Ther. 2020 Dec;9(4):785-796. doi: 10.1007/s40121-020-00311-8. Epub 2020 Jul 24. PMID 32710245
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112266 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject who was not able to come at Year (Y) 16 entered the study at Y17. At Y16, 1 subject was administered a challenge dose of Engerix-B vaccine and at Y18 and Y20, 2 subjects were administered a challenge dose of Havrix vaccine. None of the subjects received a challenge dose at Y17 and Y19.
Groups:
- Twinrix Group: Subjects who received 3 doses of Twinrix (lot A, B or C) in the primary study.
  As lot to lot consistency was assessed during the primary study, the 3 groups (lot A, B or C) were pooled into the Twinrix Group for data analyses during the first long-term follow-up NCT00289718 and this long-term follow-up.
  A challenge dose of the Havrix or Engerix-B vaccines can be administered in this study based on serology results at each time point.
Period: Year 16
Arm/Group | Twinrix Group
Started | 49
Completed | 49
Not Completed | 0
Period: Year 17
Arm/Group | Twinrix Group
Started | 48
Completed | 48
Not Completed | 0
Period: Year 18
Arm/Group | Twinrix Group
Started | 44
Completed | 44
Not Completed | 0
Period: Year 19
Arm/Group | Twinrix Group
Started | 45
Completed | 45
Not Completed | 0
Period: Year 20
Arm/Group | Twinrix Group
Started | 45
Completed | 44 (One subject returned at Y20 but did not do lab test because subject met a study exclusion criteria.)
Not Completed | 1
Not completed — Others | 1

BASELINE CHARACTERISTICS:
Arm/Group | Twinrix Group
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 16 Population: Number of participants at year 16 are equal to the overall number of participants analyzed, which represents the highest number of participants from year 16 to year 20.
  Years | 37.4 (5.66)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 17 Population: Number of participants analyzed represents all subjects who returned at the year 17 annual time point.
  Years
    number analyzed (Participants) | 48
    (all) | 38.6 (5.73)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 18 Population: Number of participants analyzed represents all subjects who returned at the year 18 annual time point.
  Years
    number analyzed (Participants) | 44
    (all) | 39.7 (5.89)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 19 Population: Number of participants analyzed represents all subjects who returned at the year 19 annual time point.
  Years
    number analyzed (Participants) | 45
    (all) | 40.7 (5.88)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 20 Population: Number of participants analyzed represents all subjects who returned at the year 20 annual time point.
  Years
    number analyzed (Participants) | 45
    (all) | 41.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 16 Population: Number of participants at year 16 are equal to the overall number of participants analyzed, which represents the highest number of participants from year 16 to year 20.
  Participants
    Female | 40
    Male | 9
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 17 Population: Number of participants analyzed represents all subjects who returned at the year 17 annual time point.
  Participants
    number analyzed (Participants) | 48
    Female | 38
    Male | 10
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 18 Population: Number of participants analyzed represents all subjects who returned at the year 18 annual time point.
  Participants
    number analyzed (Participants) | 44
    Female | 35
    Male | 9
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 19 Population: Number of participants analyzed represents all subjects who returned at the year 19 annual time point.
  Participants
    number analyzed (Participants) | 45
    Female | 36
    Male | 9
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 20 Population: Number of participants analyzed represents all subjects who returned at the year 20 annual time point.
  Participants
    number analyzed (Participants) | 45
    Female | 36
    Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seropositive for Anti-hepatitis A Virus Antibodies (Anti-HAV) and Anti-hepatitis B Surface Antigen (Anti-HBs) Antibodies and With Anti-HBs Antibody Concentrations >= 10 Milliinternational Units Per Milliliter (mIU/mL)
Description: Seropositivity for anti-HAV antibodies is defined as antibody concentrations >= 15 milliinternational units per milliliter (mIU/mL). Seropositivity for anti-HBs antibodies is defined as antibody concentrations >= 6.2 mIU/mL.
Time Frame: At Years 16, 17, 18, 19 and 20.
Population: The analysis was performed on the long-term according-to-protocol (LT ATP) cohort for immunogenicity which included subjects who returned at a particular blood sampling time point, who were included in the ATP analysis for the primary study and who did not receive hepatitis A or B vaccination that was not specified in the protocol.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 28
Subjects
  anti-HAV >= 15 mIU/mL [at Year 16] (N=28) | 28
  anti-HBs >= 6.2 mIU/mL [at Year 16] (N=28) | 27
  anti-HBs >= 10 mIU/mL [at Year 16] (N=28) | 27
  anti-HAV >= 15 mIU/mL [at Year 17] (N=27) | 26
  anti-HBs >= 6.2 mIU/mL [at Year 17] (N=27) | 25
  anti-HBs >= 10 mIU/mL [at Year 17] (N=27) | 25
  anti-HAV >= 15 mIU/mL [at Year 18] (N=25) | 25
  anti-HBs >= 6.2 mIU/mL [at Year 18] (N=25) | 23
  anti-HBs >= 10 mIU/mL [at Year 18] (N=25) | 23
  anti-HAV >= 15 mIU/mL [at Year 19] (N=25) | 24
  anti-HBs >= 6.2 mIU/mL [at Year 19] (N=25) | 23
  anti-HBs >= 10 mIU/mL [at Year 19] (N=25) | 23
  anti-HAV >= 15 mIU/mL [at Year 20] (N=25) | 24
  anti-HBs >= 6.2 mIU/mL [at Year 20] (N=25) | 23
  anti-HBs >= 10 mIU/mL [at Year 20] (N=25) | 23

2. Primary Outcome: Anti-HAV and Anti-HBs Geometric Mean Concentrations (GMCs)
Description: Concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Years 16, 17, 18, 19 and 20.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 28
mIU/mL
  anti-HAV [at Year 16] (N=28) | 262.5 [189.9 to 362.9]
  anti-HBs [at Year 16] (N=28) | 79.9 [45.2 to 141.0]
  anti-HAV [at Year 17] (N=27) | 369.4 [257.9 to 529.1]
  anti-HBs [at Year 17] (N=27) | 71.7 [39.6 to 129.8]
  anti-HAV [at Year 18] (N=25) | 237.7 [163.7 to 345.4]
  anti-HBs [at Year 18] (N=25) | 61.3 [36.8 to 102.3]
  anti-HAV [at Year 19] (N=25) | 234.3 [159.0 to 345.5]
  anti-HBs [at Year 19] (N=25) | 59.7 [35.1 to 101.4]
  anti-HAV [at Year 20] (N=25) | 229.3 [157.1 to 334.6]
  anti-HBs [at Year 20] (N=25) | 57.7 [33.6 to 99.1]

3. Secondary Outcome: Anti-HBs Concentrations After the Challenge Dose of Engerix-B
Description: Concentration was given in mIU/mL.
  Only 1 subject was eligible for the challenge dose of Engerix-B at the Year 16 time point. Therefore the values for this subject are given without a measure of dispersion.
Time Frame: Before, 14 days and one month (30 days) after the challenge dose of Engerix-B.
Population: The analysis was performed on the long-term according-to-protocol (LT ATP) cohort for immunogenicity which included subjects who returned at the blood sampling time point for whom results were available and who received a challenge dose of Engerix-B vaccine because their anti-HBs antibody concentrations were < 10 mIU/mL.
Measure: Number; unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
mIU/mL
  before challenge dose at Year 16 | 7.86
  14 days after challenge dose at Year 16 | 50640.0
  1 month (Day 30) after challenge dose at Year 16 | 31442.0

4. Secondary Outcome: Anti-HAV Concentrations After the Challenge Dose of Havrix
Description: Concentration was given in mIU/mL. Only 2 subjects were eligible for the challenge dose of Havrix, one at Year 18 and another at Year 20 time point. Therefore the values for these subject are given without a measure of dispersion.
Time Frame: Before, 14 days and one month (30 days) after the challenge dose of Havrix.
Population: The analysis was performed on the long-term according-to-protocol (LT ATP) cohort for immunogenicity which included subjects who returned at the blood sampling time point for whom results were available and who received a challenge dose of Havrix vaccine because their anti-HAV antibody concentrations were < 15 mIU/mL.
Measure: Number; unit: mIU/mL
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
mIU/mL
  before challenge dose at Year 18 | 25
  14 days after challenge dose at Year 18 | 3421
  1 month (Day 30) after challenge dose at Year 18 | 3389
  before challenge dose at Year 20 | 19
  14 days after challenge dose at Year 20 | 1096
  1 month (Day 30) after challenge dose at Year 20 | 1060

5. Secondary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose of Engerix-B
Description: At Year 16 only 1 subject was eligible for the challenge dose of Engerix-B.
  Anti-HBs anamnestic response to the challenge dose was defined as:
  * Anti-HBs antibody concentrations >= 10 mIU/mL at one month post-challenge dose in subjects seronegative at the pre-challenge time point.
  * At least a 4-fold increase in anti-HBs antibody concentrations, at one month post-challenge dose in subjects seropositive at the pre-challenge time point.
Time Frame: 30 days after the challenge dose of Engerix-B.
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects | 1

6. Secondary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose of Havrix
Description: Anti-HAV anamnestic response to the challenge dose was defined as:
  * Anti-HAV antibody concentrations ≥ 15 mIU/mL at one month post-challenge dose, in subjects seronegative at the pre-challenge time point.
  * At least a 2-fold increase in anti-HAV antibody concentrations one month after the challenge dose, in subjects having anti-HAV antibody concentrations ≥ 100 mIU/mL at the pre-challenge time point.
  * Or at least a 4-fold increase in anti-HAV antibody concentrations one month after the challenge dose, in seropositive subjects having anti-HAV antibody concentrations < 100 mIU/mL at the pre-challenge time-point.
Time Frame: 30 days after the challenge dose of Havrix.
Population: as for outcome 4
Measure: Number; unit: subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
subjects | 2

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: At Year 16, 1 subject was administered a challenge dose of Engerix-B and at Y18 and Y20, 2 subjects were administered a challenge dose of Havrix.
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: 31 days (Days 0-30) after the challenge dose of Engerix-B and Havrix.
Population: The analysis was performed on the long-term total cohort which included subjects who returned at the blood sampling time point for whom results were available and who received a challenge dose of Engerix-B vaccine or Havrix.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 3
Subjects | 1

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Only 1 subject received a challenge dose at Year 16 of Engerix-B.
  An SAE is any untoward medical occurrence that: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 31-day (Days 0-30) follow-up period after the Engerix-B challenge dose.
Population: The analysis was performed on the long-term total cohort which included subjects who returned at the blood sampling time point for whom results were available and who received a challenge dose of Engerix-B vaccine because their anti-HBs antibody concentrations were < 10 mIU/mL.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 1
Subjects | 0

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: One subject received a challenge dose of Havrix at Year 18 and another at Year 20.
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the 31-day (Days 0-30) follow-up period after the Havrix challenge dose.
Population: The analysis was performed on the long-term total cohort which included subjects who returned at the blood sampling time point for whom results were available and who received a challenge dose of Havrix vaccine because their anti-HAV antibody concentrations were < 15 mIU/mL.
Measure: Number; unit: subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 2
subjects | 0

10. Secondary Outcome: Number of Subjects Reporting SAEs Related to Study Participation or a Concurrent GSK Medication
Description: An SAE is any untoward medical occurrence that: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Up to Year 20.
Population: The LT Total cohort included all subjects who returned at each annual time point and who belonged to the Total cohort in the primary study.
Measure: Number; unit: Subjects
Arm/Group | Twinrix Group
Number analyzed (Participants) | 49
Subjects | 0

ADVERSE EVENTS:
Time Frame: SAEs: During the 31-day (Days 0 to 30) follow-up period after the challenge dose and from the beginning of the long term follow-up to Year 20; Unsolicited symptoms: During the 31-day (Days 0 to 30) follow-up period after the challenge dose.
Description: As no challenge dose was administered during Years 17 and 19 time points, SAEs and other adverse events were not assessed. At Year 16, 1 subject was administered a challenge dose of Engerix-B vaccine and at Years 18 and 20, 2 subjects were administered a challenge dose of Havrix vaccine, for whom the SAEs and other adverse events were assessed during the 31 day period post challenge dose. SAEs were also collected for the entire safety follow-up.
Arm/Group | Twinrix Group
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Twinrix Group (N=3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A decrease in specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody(10-100 mIU/mL).The tables show updated results following complete retesting/reanalysis for Y16-18.Y19 & 20 results were only analyzed by CLIA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.